CLINICAL TRIAL: NCT01435733
Title: Parenting a Child With Autism Spectrum Disorder and Marital Status
Status: Suspended | Type: Observational
Why Stopped: Recruitment Status
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-11-8552-LG-CTIL
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Divorce
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parents of children with ASD: Parents with one or more children diagnosed with Autism Spectrum Disorder

SUMMARY:
The purpose of this study is to investigate whether the presence of a child with Autism Spectrum Disorder places parents at increased risk for divorce.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) are lifelong neurodevelopmental disorders involving a triad of impairments in communication and social reciprocity and increases in repetitive/restricted interests and behaviors. ASD includes: autistic disorder, Asperger's syndrome, pervasive developmental disorder not otherwise specified (PDD-NOS), Rett's syndrome, and childhood disintegrative disorder as pervasive developmental disorders (American Psychiatric Association [DSM-IV-TR], 2000).

Few disabilities appear to be more taxing on parents than ASDs.Parents of children with ASD fare worse on a variety of measures of well-being than parents of children without disabilities as well as parents of children with other types of disabilities.

Studies investigating the impact of a child with disabilities, specifically ASD, are inconclusive. However, parents of children with ASD may be at increased risk for divorce due to a variety of personal and disability related factors. In Israel the relationship of having a child with autism on the probability of divorce has not been tested yet. The aim of this study is to profile this relationship and determine the magnitude and directionality of the effect raising ASD children has on the resilience of the institution of marriage and the satisfaction both partners derive. This will be tested using a short telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* parents to a child with ASD

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Couples who have children with ASD will be recruited to participate in this study from the Weinberg Child Development Center in the Edmond and LilySafra Children'shospital, ShebaMedical Center, Ramat-Gan, Israel. Parents will be contacted through the telephone and provided with a brief explanation about the study. Participation will be voluntary with no monetary compensation. Parents who volunteer to participate will then be presented with a short telephone survey, asking them about their marital status and other variables related to the link between parenting an ASD child and their marital status.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-09-01; Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
lower or higher levels of divorce | not relevant (phone survey)
  lower or higher levels of divorce

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center; Gilad Gal, Ph.D, Principal Investigator — Tel Aviv-Yafo Academic College; Klara Zislin, BA, Study Director — Sheba Medical Center
Locations (1):
- Weinberg Child Development Center, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No